CLINICAL TRIAL: NCT02072603
Title: Evaluation of the HITSystem to Improve Early Infant Diagnosis Outcomes in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Kessler, PhD, MPH (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Sarah Kessler, PhD, MPH, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13793; 1R01HD076673-01A1 (NIH)
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: HIV
Keywords: Infant HIV; Kenya; HITSystem; EID care; Early Infant Diagnosis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Hospitals (Experimental): HITSystem implementation at hospital and its affiliated laboratory
  Interventions: Other: HITSystem
- Control Hospitals (Active Comparator): Existing standard of EID care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: HITSystem — Online, automated program designed to overcome current EID barriers by providing efficient prospective tracking of HIV-exposed infants and triggering electronic action "alerts" for both EID providers and lab technicians when time sensitive interventions are overdue for specific infants.
  Other Names: HIV Infant Tracking System
  Arms: Intervention Hospitals
Other: Standard of Care — current procedures that follow Kenyan National EID guidelines to diagnose and manage HIV infection among HIV-exposed infants.
  Arms: Control Hospitals

SUMMARY:
The purpose of this study is to determine the effectiveness of the HITSystem in maximizing early infant diagnosis (EID) service utilization for HIV-exposed infants and early antiretroviral therapy (ART) initiation for infants diagnosed with HIV.

DETAILED DESCRIPTION:
The current EID system is hampered by significant structural barriers that contribute to late and sporadic testing of HIV-exposed infants, lost or delayed test results from the laboratory, and the absence of a reliable system to notify mothers of test results or the need to return to the hospital.

Consequently, in Kenya only about one-third of HIV-exposed infants receive complete EID care through 18 months of age, and less than 20% of diagnosed HIV+ infants are initiated on life saving ART.

To maximize both the benefits and efficiencies of EID efforts, the investigators have developed a system strengthening intervention called the HIV Infant Tracking System (HITSystem©). The HITSystem intervention is an online, automated intervention designed to overcome current EID barriers by providing efficient prospective tracking of HIV- exposed infants and triggering electronic action 'alerts' for both EID providers and lab technicians when time sensitive interventions are overdue for specific infants. A built-in text messaging system sends text messages to mothers' cell phones when test results are ready or follow up visits are needed. The ultimate goals of the HITSystem are to maximize (a) EID service utilization for HIV-exposed infants (retention until 18 months) and (b) early ART initiation for infants diagnosed HIV+, by facilitating collaboration and accountability between key stakeholders (hospitals, laboratories and mothers) to improve EID outcomes.

Our pilot data from two hospitals in Kenya (one urban, one peri-urban) demonstrate the acceptability and feasibility of implementing this intervention. Using a pre-post intervention design the investigators compared EID outcomes from n=330 mother-infant pairs assessed by retrospective chart review during the 12 months prior to the initiation of the intervention to n=460 mother-infant pairs enrolled in the HITSystem intervention over the course of several months (9 and 6 months, respectively). Pilot data indicate a 3 fold increase in EID retention (31% vs. 97%, p<0.001), and more than doubled infant ART initiation rates (44% vs. 95%, p<0.001).14 These data have resulted in great interest and support from the Kenya Ministry of Health for this study, the findings of which will influence national EID dissemination decisions.

To more rigorously evaluate the impact of the HITSystem intervention on EID care in a low-resource country and implications for the feasibility of scaling up this intervention, the investigators will use a cluster randomized control trial among 6 Kenyan government hospitals (3 intervention and 3 standard of care; matched). Three specific aims guide the proposed study:

Aim 1. Conduct a randomized controlled trial to evaluate the efficacy of the HITSystem in improving the timely provision of 8 critical intervention benchmarks for optimal Early Infant Diagnosis of HIV and management.

Aim 2. To identify among HIV-exposed infants predictors of (1) incomplete EID care and (2) time periods most vulnerable to loss of contact at both intervention and control sites.

Aim 3. To estimate the incremental cost-effectiveness of the HITSystem in improving complete EID care across study arms, and to assess user satisfaction among key stakeholders.

This study will scientifically evaluate the public health impact of the HITSystem to improve critical EID outcomes in low-resource settings. Cost-effectiveness analyses will inform the feasibility of scaling up the HITSystem in other settings, and opportunities to adapt the technology to address other health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ mother whose infant is <18 months of age
* Ability to provide consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1815 (Actual)
Dates: Start 2014-03-30 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Complete EID Retention | 18 months
  An aggregate measure of complete EID retention will be calculated (y/n) for each infant. Complete EID retention indicates the infant received all indicated services along the EID cascade as detailed below in the 8 critical interventions for EID of HIV. The proportion of HIV-exposed infants with complete EID retention will be compared between groups.
  1. Initiation of OI prophylaxis.
  2. Collect dried blood spot (DBS) for PCR test.
  3. Receipt of DBS at lab.
  4. Return of PCR results from lab.
  5. Notify mother of PCR results.
  6. Initiate all HIV-infected infants on ART.
  7. Retest all HIV-negative infants at 9 m, initiate ART if applicable.
  8. Retest all HIV-negative infants at 18 ms, initiate ART if applicable

SECONDARY OUTCOMES:
Efficiency of EID testing and notification cycle | 18 months
  Measuring turn-around time for the complete testing and notification cycle i.e, from sample collection to notifying mothers of results. Measured in number of weeks.
Rapid treatment initiation among HIV+ infants | 18 months
  Time from notifying mother of HIV+ test result and initiating infant on ART, measured in days
Mother-to-child transmission of HIV occurring between first and follow up tests | 18 months
  Mother-to-child transmission of HIV occurring between first and follow up tests, e.g. infants who are uninfected at first test (6 wks) but test positive at either the 9 or 18 month follow up test
Cost effectiveness of HITSystem | 18 months
  Intervention costs per outcome achieved using the HITSystem versus the standard of care control condition. Savings resulting from HITSystem use will also be measured.
Infant Mortality | 18 months
  Document the number of infants enrolled in EID who die before the end of the study period. Cause of death will be recorded.
Infant age at ART initiation | 18 months
  The age at which an HIV+ infant was initiated on ART
Optimal EID Index | 18 months
  To calculate a score for the Optimal EID Index, the infant will receive a score for each of the 8 EID interventions for which they were eligible; if it was completed (1-point) or never completed (0 points) and whether it was completed on-time (1 point) or off-time (0 points) for a maximum score of 16 and a minimum score of 0.
  1. Initiation of OI prophylaxis at 6 wks.
  2. Collect dried blood spot (DBS) for PCR test by 6 wks.
  3. Receipt of DBS at lab within 10 days of collection.
  4. Return of PCR results from lab within 2 wks.
  5. Notify mother within 2 wks of the EID provider receiving results.
  6. Initiate all HIV-infected infants on ART w/in 4 weeks of notifying the mother.
  7. Retest all HIV-negative infants at 9 m, initiate ART w/in 4 wks if applicable.
  8. Retest all HIV-negative infants at 18 ms, initiate ART w/in 4 wks if applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah F Kessler, PhD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (2):
- University of Kansas Medical Center, Kansas City, Kansas, United States
- Kenyan Medical Research Institute, Nairobi, Kenya

REFERENCES:
- [Background] Finocchario-Kessler S, Goggin K, Khamadi S, Gautney B, Dariotis JK, Bawcom C, Cheng AL, Nazir N, Martin C, Ruff A, Sweat M, Okoth V. Improving early infant HIV diagnosis in Kenya: study protocol of a cluster-randomized efficacy trial of the HITSystem. Implement Sci. 2015 Jul 9;10:96. doi: 10.1186/s13012-015-0284-3. PMID 26155932
- [Background] Finocchario-Kessler S, Gautney BJ, Khamadi S, Okoth V, Goggin K, Spinler JK, Mwangi A, Kimanga D, Clark KF, Olungae HD, Preidis GA; HITSystem Team. If you text them, they will come: using the HIV infant tracking system to improve early infant diagnosis quality and retention in Kenya. AIDS. 2014 Jul;28 Suppl 3(0 3):S313-21. doi: 10.1097/QAD.0000000000000332. PMID 24991904
- [Result] Goggin K, Wexler C, Nazir N, Staggs VS, Gautney B, Okoth V, Khamadi SA, Ruff A, Sweat M, Cheng AL, Finocchario-Kessler S. Predictors of Infant Age at Enrollment in Early Infant Diagnosis Services in Kenya. AIDS Behav. 2016 Sep;20(9):2141-50. doi: 10.1007/s10461-016-1404-z. PMID 27108002
- [Result] Wexler C, Brown M, Hurley EA, Ochieng M, Goggin K, Gautney B, Maloba M, Lwembe R, Khamadi S, Finocchario-Kessler S. Implementing eHealth Technology to Address Gaps in Early Infant Diagnosis Services: Qualitative Assessment of Kenyan Provider Experiences. JMIR Mhealth Uhealth. 2018 Aug 22;6(8):e169. doi: 10.2196/mhealth.9725. PMID 30135052
- [Result] Finocchario-Kessler S, Gautney B, Cheng A, Wexler C, Maloba M, Nazir N, Khamadi S, Lwembe R, Brown M, Odeny TA, Dariotis JK, Sandbulte M, Mabachi N, Goggin K. Evaluation of the HIV Infant Tracking System (HITSystem) to optimise quality and efficiency of early infant diagnosis: a cluster-randomised trial in Kenya. Lancet HIV. 2018 Dec;5(12):e696-e705. doi: 10.1016/S2352-3018(18)30245-5. Epub 2018 Oct 8. PMID 30309787
- [Result] Brown M, Wexler C, Gautney B, Goggin K, Hurley EA, Odeny B, Maloba M, Lwembe R, Sandbulte M, Finocchario-Kessler S. eHealth Interventions for Early Infant Diagnosis: Mothers' Satisfaction with the HIV Infant Tracking System in Kenya. AIDS Behav. 2019 Nov;23(11):3093-3102. doi: 10.1007/s10461-019-02579-5. PMID 31313093
- [Result] Goggin K, Hurley EA, Staggs VS, Wexler C, Nazir N, Gautney B, Khamadi SA, Maloba M, Lwembe R, Finocchario-Kessler S. Rates and Predictors of HIV-Exposed Infants Lost to Follow-Up During Early Infant Diagnosis Services in Kenya. AIDS Patient Care STDS. 2019 Aug;33(8):346-353. doi: 10.1089/apc.2019.0050. PMID 31369296
- [Result] Wexler C, Nazir N, Gautney B, Maloba M, Brown M, Goggin K, Lwembe R, Finocchario-Kessler S. Predictors of Early ART Initiation Among HIV + Infants in Kenya: A Retrospective Review of HITSystem Data from 2013 to 2017. Matern Child Health J. 2020 Jun;24(6):739-747. doi: 10.1007/s10995-020-02909-3. PMID 32285335
- [Result] Hurley EA, Odeny B, Wexler C, Brown M, MacKenzie A, Goggin K, Maloba M, Gautney B, Finocchario-Kessler S. "It was my obligation as mother": 18-Month completion of Early Infant Diagnosis as identity control for mothers living with HIV in Kenya. Soc Sci Med. 2020 Apr;250:112866. doi: 10.1016/j.socscimed.2020.112866. Epub 2020 Feb 27. PMID 32145483